CLINICAL TRIAL: NCT06744205
Title: A Phase I/II, Randomized, Modified Double-blind Study to Investigate the Safety and Immunogenicity of Different Doses of Hexavalent Influenza mRNA HA + mRNA NA Vaccine in Adult Participants 50 Years of Age and Older
Brief Title: A Study on the Safety and Immunogenicity of Hexavalent Influenza mRNA Vaccine in Adult Participants 50 Years of Age and Older
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FBP00021; U1111-1303-3537 (Registry Identifier: WHO ICTRP)
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Influenza; Healthy Volunteers
Keywords: influenza, flu, vaccine, hexavalent
MeSH Terms: conditions — Influenza, Human | interventions — RNA, Messenger; Hemagglutinins; Vaccines; Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Dose escalation with sequential enrollment of sentinel cohorts followed by parallel enrollment of the main cohort.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Modified double-blind (participants; sites, except for those preparing/administering study intervention; and Sponsor will be blinded. Sponsor's internal safety monitoring team could be unblinded if necessary)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Group 1 - Hexavalent (Combination 1) (Experimental): Participants will receive single dose of hexavalent influenza mRNA vaccine composed of differing dose levels of TIV mRNA-HA Vaccine 1 in combination with TIV mRNA-NA (Combination 1)
  Interventions: Biological: Trivalent (TIV) messenger ribonucleic acid (mRNA) hemagglutinin (HA) Vaccine 1; Biological: TIV mRNA-neuraminidase (NA)
- Group 2 - Hexavalent (Combination 2) (Experimental): Participants will receive single dose of hexavalent influenza mRNA vaccine composed of differing dose levels of TIV mRNA-HA Vaccine 1 in combination with TIV mRNA-NA (Combination 2)
  Interventions: Biological: Trivalent (TIV) messenger ribonucleic acid (mRNA) hemagglutinin (HA) Vaccine 1; Biological: TIV mRNA-neuraminidase (NA)
- Group 3 - Hexavalent (Combination 3) (Experimental): Participants will receive single dose of hexavalent influenza mRNA vaccine composed of differing dose levels of TIV mRNA-HA Vaccine 1 in combination with TIV mRNA-NA (Combination 3)
  Interventions: Biological: Trivalent (TIV) messenger ribonucleic acid (mRNA) hemagglutinin (HA) Vaccine 1; Biological: TIV mRNA-neuraminidase (NA)
- Group 4 - Hexavalent (Combination 4) (Experimental): Participants will receive single dose of hexavalent influenza mRNA vaccine composed of differing dose levels of TIV mRNA-HA Vaccine 1 in combination with TIV mRNA-NA (Combination 4)
  Interventions: Biological: Trivalent (TIV) messenger ribonucleic acid (mRNA) hemagglutinin (HA) Vaccine 1; Biological: TIV mRNA-neuraminidase (NA)
- Group 5 - Hexavalent (Combination 5) (Experimental): Participants will receive single dose of hexavalent influenza mRNA vaccine composed of differing dose levels of TIV mRNA-HA Vaccine 1 in combination with TIV mRNA-NA (Combination 5)
  Interventions: Biological: Trivalent (TIV) messenger ribonucleic acid (mRNA) hemagglutinin (HA) Vaccine 1; Biological: TIV mRNA-neuraminidase (NA)
- Group 6 - Hexavalent (Combination 6) (Experimental): Participants will receive single dose of hexavalent influenza mRNA vaccine composed of differing dose levels of TIV mRNA-HA Vaccine 1 in combination with TIV mRNA-NA (Combination 6)
  Interventions: Biological: Trivalent (TIV) messenger ribonucleic acid (mRNA) hemagglutinin (HA) Vaccine 1; Biological: TIV mRNA-neuraminidase (NA)
- Group 7 - TIV mRNA-HA Vaccine 1 (Experimental): Participants will receive a single dose of TIV mRNA-HA Vaccine 1
  Interventions: Biological: Trivalent (TIV) messenger ribonucleic acid (mRNA) hemagglutinin (HA) Vaccine 1
- Group 8 - TIV mRNA-NA (Experimental): Participants will receive a single dose of TIV mRNA-NA
  Interventions: Biological: TIV mRNA-neuraminidase (NA)
- Group 9 - TIV mRNA-HA Vaccine 2 (Experimental): Participants will receive single dose of TIV mRNA-HA Vaccine 2
  Interventions: Biological: TIV mRNA-HA Vaccine 2
- Group 10 - QIV-SD (Active Comparator): Participants will receive single dose of QIV-SD vaccine (for participants 50 to 64 years of age only)
  Interventions: Biological: Quadrivalent Influenza Standard Dose Vaccine
- Group 11 - QIV-HD (Active Comparator): Participants will receive single dose of QIV-HD vaccine
  Interventions: Biological: Quadrivalent Influenza Vaccine High Dose

INTERVENTIONS:
Biological: Trivalent (TIV) messenger ribonucleic acid (mRNA) hemagglutinin (HA) Vaccine 1 — * Pharmaceutical form: solution for injection in a vial
  * Route of administration: Intramuscular injection
  Arms: Group 1 - Hexavalent (Combination 1); Group 2 - Hexavalent (Combination 2); Group 3 - Hexavalent (Combination 3); Group 4 - Hexavalent (Combination 4); Group 5 - Hexavalent (Combination 5); Group 6 - Hexavalent (Combination 6); Group 7 - TIV mRNA-HA Vaccine 1
Biological: TIV mRNA-neuraminidase (NA) — * Pharmaceutical form: solution for injection in a vial
  * Route of administration: Intramuscular injection
  Arms: Group 1 - Hexavalent (Combination 1); Group 2 - Hexavalent (Combination 2); Group 3 - Hexavalent (Combination 3); Group 4 - Hexavalent (Combination 4); Group 5 - Hexavalent (Combination 5); Group 6 - Hexavalent (Combination 6); Group 8 - TIV mRNA-NA
Biological: TIV mRNA-HA Vaccine 2 — * Pharmaceutical form: solution for injection in a vial
  * Route of administration: Intramuscular injection
  Arms: Group 9 - TIV mRNA-HA Vaccine 2
Biological: Quadrivalent Influenza Standard Dose Vaccine — * Pharmaceutical form: Liquid suspension for injection in pre-filled syringe
  * Route of administration: Intramuscular injection
  Other Names: Fluzone Qudrivalent®
  Arms: Group 10 - QIV-SD
Biological: Quadrivalent Influenza Vaccine High Dose — * Pharmaceutical form: Liquid suspension for injection in pre-filled syringe
  * Route of administration: Intramuscular injection
  Other Names: Fluzone High-Dose Quadrivalent®
  Arms: Group 11 - QIV-HD

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a single intramuscular injection of different formulations of a hexavalent influenza messenger ribonucleic acid (mRNA) vaccine composed of differing dose levels of trivalent (TIV) mRNA hemagglutinin (HA) in combination with TIV mRNA-neuraminidase (NA) compared to an active control ((Fluzone standard-dose quadrivalent influenza vaccine (QIV-SD) or Fluzone high-dose quadrivalent influenza vaccine (QIV-HD) in adults 50 years of age and older.

DETAILED DESCRIPTION:
Study details include the following:

* Study Duration: approximately 12 months for each participant
* Treatment: 1 injection of hexavalent vaccine, trivalent vaccine, or active control
* Visit frequency: Day (D) 01, D03, D09, D29, and D181; D366 (telephone call)
* Dose escalation with sequential enrollment of sentinel cohorts followed by parallel enrollment of the main cohort

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 50 years on the day of inclusion
* A female participant is eligible to participate if she is not pregnant or breastfeeding and one of the following conditions applies:

  * Is of non-childbearing potential. To be considered of non-childbearing potential, a female must be postmenopausal for at least 1 year, or surgically sterile.

OR

* Is of childbearing potential and agrees to use an effective contraceptive method or abstinence from at least 4 weeks prior to study intervention administration until at least 12 weeks after study intervention administration.

A female participant of childbearing potential must have a negative highly sensitive pregnancy test (urine or serum as required by local regulation) within 8 hours prior to administration of study intervention.

Exclusion Criteria:

Participants are not eligible for the study if any of the following criteria are met:

* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the study intervention components (eg, polyethylene glycol, polysorbate); history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances; any allergic reaction (eg, anaphylaxis) after administration of mRNA vaccine
* Previous history of myocarditis, pericarditis, and/or myopericarditis
* Known history of previous episodes of Guillain-Barré syndrome, neuritis (including Bell's palsy), convulsions, encephalitis, transverse myelitis, and vasculitis
* Participants with an electrocardiogram that is consistent with possible myocarditis or pericarditis or, in the opinion of the investigator, demonstrates clinically relevant abnormalities that may affect participant safety or study results
* Self-reported thrombocytopenia, contraindicating intramuscular (IM) vaccination based on Investigator's judgment
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination based on Investigator's judgment
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness / infection (according to investigator's judgement) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of vaccination. A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Alcohol, prescription drug, or substance abuse that, in the opinion of the Investigator, might interfere with the study conduct or completion
* Participant who had acute infectious symptoms or a positive SARS-CoV-2 RT-PCR or antigen test in the past 10 days prior to the first visit (V01)
* Receipt of any vaccine in the 4 weeks preceding study intervention administration or planned receipt of any vaccine in the 4 weeks following study intervention administration
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Previous vaccination against influenza in the previous 6 months with an investigational or marketed vaccine
* Receipt of any mRNA vaccine/product in the 2 months preceding study intervention administration or planned receipt of any mRNA vaccine in the 2 months after study vaccination
* Participation at the time of study enrollment (or in the 4 weeks preceding study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure
* Self-reported or documented seropositivity for human immunodeficiency virus, hepatitis B virus, or hepatitis C virus

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1162 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-04-16 (Estimated); Study Completion 2026-04-16 (Estimated)

PRIMARY OUTCOMES:
Number of participants with immediate unsolicited systemic adverse events (AEs) | Within 30 minutes after injection
  Unsolicited systemic AEs that occur within 30 minutes after vaccination
Number of participants with solicited injection site reactions | Up to 7 days after injection
  Solicited injection site reactions pre-listed in the participant diary and in the case report form CRF
Number of participants with solicited systemic reactions | Up to 7 days after injection
  Solicited systemic reactions pre-listed in the participant diary and in the CRF
Number of participants with unsolicited AEs | Up to 28 days after injection
  AEs that do not fulfill the conditions of solicited reactions
Number of participants with medically attended adverse events (MAAEs) | Up to 180 days after injection
  MAAEs reported up to 180 days after injection
Number of participants with serious adverse events (SAEs) | SAEs throughout the study (Up to approximately 12 months)
  Throughout the study
Number of participants with adverse events of special interest (AESIs) | AESIs throughout the study (Up to approximately 12 months)
  Throughout the study
Number of participants with out-of-range biological test results | Up to 8 days after injection
  Out-of-range biological test results (including shift from baseline values)
Hemagglutinin inhibition (HAI) titers | At Day 1 and Day 29
  HAI titers at D01 and D29
Individual HAI antibody (Ab) titer ratio D29/D01 | At Day 1 and Day 29
  Individual HAI Ab titer ratio D29/D01
Seroconversion (HAI Ab titer) | At Day 1 and Day 29
  Number of participants with HAI Ab titer < 10 [1/dil] at Day 1 and post-injection titer ≥ 40 [1/dil] at Day 29, or titer ≥ 10 [1/dil] at Day 1 and a ≥ 4-fold increase in titer [1/dil] at Day 29
HAI Ab titer ≥ 40 (1/dil) | At Day 29
  HAI Ab titer ≥ 40 (1/dil) at D29
Neuraminidase inhibition (NAI) titers | At Day 1 and Day 29
  NAI titers at D01 and D29
Individual NAI Ab titer ratio D29/D01 | At Day 1 and Day 29
  Individual NAI Ab titer ratio D29/D01
Seroconversion (NAI Ab titer) | At Day 1 and Day 29
  Number of participants with NAI Ab titer < 10 [1/dil] at D01 and post-injection titer ≥ 40 [1/dil] at D29, or titer ≥ 10 [1/dil] at D01 and a ≥ 4-fold increase in titer [1/dil] at D29)
NAI Ab titer ≥ 40 (1/dil) | At Day 29
  NAI Ab titer ≥ 40 (1/dil) at D29
2-fold and 4-fold rise in NAI titers | Day 1 to Day 29
  2-fold and 4-fold rise in NAI titers from D01 to D29

SECONDARY OUTCOMES:
Neutralizing antibodies titers | At Day 1 and Day 29
  Neutralizing antibodies titers at D01 and D29
Individual neutralizing antibodies titer ratio | At Day 1 and Day 29
  Individual neutralizing antibodies titer ratio D29/D01
2-fold and 4-fold increase in neutralizing titers | Day 1 to Day 29
  2-fold and 4-fold increase in neutralizing titers D01 through D29

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (24):
- United States (21):
  - Accel Research Sites Network - Birmingham- Site Number : 8400008, Birmingham, Alabama
  - AMR Mobile- Site Number : 8400022, Mobile, Alabama
  - Alliance for Multispeciality Research - Clinical Research Consortium- Site Number : 8400015, Tempe, Arizona
  - AMR Miami- Site Number : 8400021, Coral Gables, Florida
  - Accel Research Sites Network - DeLand Clinical Research Unit- Site Number : 8400003, DeLand, Florida
  - Alliance for Multispeciality Research - Fort Myers- Site Number : 8400013, Fort Myers, Florida
  - Accel Research Sites - Maitland- Site Number : 8400007, Maitland, Florida
  - Innovation Medical Research Center - Palmetto Bay- Site Number : 8400011, Palmetto Bay, Florida
  - Accel Research Site - NeuroStudies.net, LLC - ERN - PPDS- Site Number : 8400001, Decatur, Georgia
  - AMR - Chicago- Site Number : 8400012, Oak Brook, Illinois
  - Alliance for Multispeciality Research - Newton- Site Number : 8400020, Newton, Kansas
  - Alliance for Multispeciality Research - Wichita East- Site Number : 8400014, Wichita, Kansas
  - Alliance for Multispeciality Research - Lexington- Site Number : 8400018, Lexington, Kentucky
  - Boston Clinical Trials- Site Number : 8400009, Boston, Massachusetts
  - ActivMed Practices & Research- Site Number : 8400005, Methuen, Massachusetts
  - Quest Research Institute- Site Number : 8400010, Farmington Hills, Michigan
  - Alliance for Multispeciality Research - Kansas City- Site Number : 8400019, Kansas City, Missouri
  - AMR Las Vegas - Site Number : 8400016, Las Vegas, Nevada
  - Coastal Carolina Research Center - North Charleston- Site Number : 8400002, North Charleston, South Carolina
  - Alliance for Multispeciality Research - Knoxville- Site Number : 8400017, Knoxville, Tennessee
  - Charlottesville Medical Research- Site Number : 8400004, Charlottesville, Virginia
- Australia (3):
  - Investigational Site Number : 0360001, Botany, New South Wales
  - Investigational Site Number : 0360003, Bayswater, Victoria
  - Investigational Site Number : 0360002, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org